CLINICAL TRIAL: NCT02493985
Title: Studying Physiological and Anatomical Cerebral Effects of Carbon Dioxide and Tilt
Acronym: SPACE-COT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Space Biomedical Research Institute (Other); DLR German Aerospace Center (Other); The University of Texas Health Science Center, Houston (Other); University of Pennsylvania (Other); Harvard University (Other); University of Cologne (Other)
Responsible Party: Principal Investigator, Eric Michael Bershad, Assistant Professor of Neurology and Space Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: H-36485
Record Dates: First submitted 2015-06-27; First posted 2015-07-10 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Brain physiology; Intracranial pressure; Cognition; Cerebrovascular; Head down tilt; Space flight
MeSH Terms: interventions — Particulate Matter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atmosphere 1 - Ambient air (Active Comparator): First, the subjects will have 1 baseline day in the upright body position. This will be followed by 28 hours of head down tilt body position and ambient air at sea level, followed by 2 hour exposure of 3% carbon dioxide inhalation.
  Interventions: Other: ambient air
- Atmosphere 2 - 0.5% CO2 (Experimental): First, the subjects will have 1 baseline day in the upright body position. This will be followed by 28 hours of head down tilt body position and air with 0.5% carbon dioxide, followed by 2 hour exposure of 3% carbon dioxide inhalation.
  Interventions: Other: 0.5% CO2

INTERVENTIONS:
Other: 0.5% CO2 — The subjects will be randomized to breath 0.5% carbon dioxide during one of the -12 degree head down tilt body position periods in crossover design
  Arms: Atmosphere 2 - 0.5% CO2
Other: ambient air — The subjects will be randomized to breath ambient air during one of the -12 degree head down tilt body position periods in crossover design
  Arms: Atmosphere 1 - Ambient air

SUMMARY:
The purpose of this study is to study the effects of carbon dioxide combined with head down tilt on cerebral physiology and anatomy. This paradigm will help establish a ground-based analog for spaceflight, and also evaluate the ability of non-invasive devices to monitor brain physiology.

DETAILED DESCRIPTION:
Many of the long duration astronauts develop visual changes, associated with neuroophthalmological abnormalities suggesting elevated intracranial pressure. There is currently no suitable ground based analog to simulate these changes on Earth, or a standard methodological approach to monitoring the combined effects of head down tilt and atmospheric carbon dioxide. Given that carbon dioxide and cephalad fluid shifting are known factors in spaceflight, we sought to evaluate an approach to monitoring these effects in healthy subject in a ground based analog on Earth.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages between 30 to 55 years old
* Body Mass Index (BMI) of 20-26 kg/m2
* Weight between 65-85 kg
* Height between 158-190 cm
* Non-smoker, for at least six months before the start of the study
* VO2 max of at least 30ml/kg/min

Exclusion Criteria:

* History of intracranial pressure elevation
* History of abnormal intraocular pressure
* Ophthalmological conditions: glaucoma, retinopathy, severe cataracts, eye trauma or implants.
* History of diseases of the optic nerve
* Pre-existing corneal injury
* History of these eye surgeries: implanted lens, corneal transplant, recent (less than 6 months) LASIK surgery
* Congenital abnormalities of the anterior chamber
* Active eye infections, recent corneal abrasions, inflammation
* Intraocular pressure greater than 20 mm Hg
* Viral or bacterial eye infection Severe dry eye syndrome
* Retinal or choroidal detachment
* More than -6,0 dpr (high myopia)
* More than +5,0 dpr
* Arm or shoulder injury in the past year
* Psychiatric conditions including major depression, bipolar disorder or severe anxiety
* History of cerebrovascular disease including brain aneurysms, stroke, transient ischemic attack, brain hemorrhage, arteriovenous malformations History of brain tumor, congenital cysts, hydrocephalus, brain injury (requiring hospitalization)
* Meningitis/encephalitis
* Epilepsy
* History of severe hypertension (> 160/90 mmHg),
* Diabetes mellitus
* Coronary artery disease
* Congestive heart failure
* Ventricular or atrial arrhythmias
* Autonomic disorders (syncope, autoimmune neuropathy)
* Hepatic disease
* Renal disease
* Chronic infections including HIV, Hepatitis B or C, Lyme disease
* History of hematological disease including hemophilia, leukemia, thrombocytosis, thrombocytopenia, myelodysplastic syndrome, autoimmune disease (lupus, rheumatoid arthritis, Sjogren's syndrome)
* History of malignancy except for basal cell carcinoma
* Chronic back pain (inability to lay in bed for long periods of time)
* Conditions that would preclude MRI including severe claustrophobia, pace maker or other metallic implants or devices
* Sleep disturbances including: obstructive sleep apnea, narcolepsy, insomnia - Medications that exert cardiovascular, cerebrovascular or psychiatric function (i.e. beta blockers, calcium channel blockers, diuretics, diamox, sedatives) Drug, medication or alcohol abuse (regular consumption of more than 20-30 g alcohol/day)*
* Smoking
* VO2 max less than 30 ml/kg/min or greater than 60 ml/kg/min
* Vegetarian, vegan
* Migraine
* Previous psychiatric illness
* Hiatus hernia
* Gastro-esophageal reflux
* Diabetes mellitus
* Rheumatic illness
* Muscle or joint disorder
* Pronounced orthostatic intolerance (< 10 min standing)
* Hyperlipidaemia
* Thyroid gland disorder: deviations from normal values for TSH in plasma
* Hyper-homocysteinaemia
* Hyperuricaemia or hypouricaemia: deviations from normal values for uric acid in plasma.
* Hypercalcaemia or hypocalcaemia: deviations from normal values for calcium in plasma.
* Iron deficiency
* Vitamin D deficiency
* Baseline blood gas values deviating from the normal reference values
* Elevated risk of venous thromboembolism including deep venous thrombosis, pulmonary embolism
* Chronic back complaints
* Participation in another clinical study within the last 3 months before start of this study
* Criminal record
* Stomach sleepers
* Any other medical condition that the investigators consider a contraindication to the study procedures that would make it unsafe or confound the measurements.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral blood flow: Transcranial doppler | 24 and 48 hours from baseline measurements
  Transcranial Doppler derived measurements of mean cerebral blood flow velocity
Changes in intracranial volume | 24 and 48 hours from baseline measurements
  Cerebrotech monitor derived intracranial fluid volume changes (percentage change)
Changes in intracranial pressure | 24 and 48 hours from baseline measurements
  Vittamed ICP meter derived intracranial pressure (mmHg)
Changes in cognitive function | 24 and 48 hours from baseline measurements
  Cognition battery score (max 1000): tests multiple cognitive domains including spatial memory, psychomotor processing speed, facial emotional recognition
Changes in cerebral blood flow: cFLOW | 24 and 48 hours from baseline measurements
  cFLOW derived changes in cerebral blood flow index

SECONDARY OUTCOMES:
Tolerability of combined -12 head down tilt and 0.5% carbon dioxide | Within 48 hours from baseline
  Assess safety outcomes: tolerance of condition through duration of study and number of adverse events
Changes in intraocular pressure | 24 and 48 hours from baseline measurements
  iCare derived intraocular pressure measurements from both eyes (mmHg)
Changes in pulmonary mechanics | 24 and 48 hours from baseline measurements
  minute ventilation, respiratory rate and vital capacity
Changes in internal jugular vein volumes | 48 hours from baseline measurements
  Ultrasound derived measure of right internal jugular vein cross sectional areas
Changes in peripheral arterial vasoreactivity | 48 hours from baseline measurements
  Ultrasound Doppler Measurement of arterial diameter and flow (cm/sec) after transient cuff occlusion of brachial artery
Changes in cardiac hemodynamics | 48 hours from baseline measurements
  Assessment of cardiac output, stroke volume, heart rate, blood pressure
Changes in olfactory threshold | 24 and 48 hours from baseline measurement
  Sniffin' sticks threshold testing for phenyethyl alcohol
Changes in pulmonary gas exchange | 24 and 48 hours from baseline measurements
  changes in arterial pH and partial pressure CO2